CLINICAL TRIAL: NCT03140618
Title: The Light- and Environment Project in Psychiatric Inpatient Care
Acronym: LEPPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Västerbotten County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 3500LJUSMILJO
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Mental Ill-health; Care Environment; Light Installations
Keywords: single-system-design; mixed methods; psychiatric inpatient care; work environment; rebuilding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LEPPIC (Experimental): The light and environment project in psychiatric inpatient care
  Interventions: Other: The light and environment project in psychiatric inpatient care

INTERVENTIONS:
Other: The light and environment project in psychiatric inpatient care — Complete rebuilding of a hospital ward.
  The ward layout is remodeled and different devices and services are installed such as light, sound, and color settings, increased opportunities for physical activity, social harmony, privacy, peace, and quiet. A comfort room and a activity room will be built.

SUMMARY:
The care environment influences both patients' experiences of care as well as staff's experiences of the work environment. A radical change in physical environment is planned at a psychiatric ward, aiming at creating a care environment that supports patients' opportunities for recovery from mental ill-health and to create a better and more attractive work environment for the staff. The rebuilding involves a new ward layout and new innovations such as light installations, a comfort room and an activity room.

The study uses a single-system design to evaluate the effects of the intervention - the rebuilt ward. Both quantitative and qualitative data will be used in the evaluation. Data will be collected using questionnaires measuring dimensions of patients' well-being and experiences of the care environment, staff's experiences of work-related stress and work environment, quality of care, a device measuring physical activity, existing clinical registers and data from medical files, staff' sick leave, participant observations, and semi-structured interviews.

This evaluation study, to our knowledge the first of it's kind in Sweden, is expected to generate important knowledge of the effect of the change process that can be used at other psychiatric wards to design the inpatient care environment. In the long run, the study could lead to a better reputation of psychiatric nursing and to more attractive workplaces.

ELIGIBILITY:
Inclusion Criteria for Patients

* 18 years or older
* Admitted to the wards during either A phase, B phase and/or follow-up

Exclusion Criteria for Patients

* Does not master the Swedish language well enough to complete questionnaires and participate in interviews

Inclusion Criteria for Staff:

* Regularly employed at the ward during A and B phase and/or follow-up.

Exclusion Criteria for Staff:

* Staff employed by the hour

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Outcome Rating Scale [patients] | Changes during baseline and intervention period (measured regularly for 12 weeks)
  The Outcome Rating Scale measures self-assessed satisfaction with life on four visual-analogue scales.
Perceived stress [staff] | Changes during baseline and intervention period (measured regularly for 12 weeks)
  PSS consists of 10 items answered on a 5-point Likert scale

SECONDARY OUTCOMES:
Quality of interactions [patients] | Changes during baseline and intervention period (measured regularly for 12 weeks)
  This is measured using The Caring Professional Scale (CPS) that consists of 14 items answered on a 5-point Likert scale.
Anxiety and depressive symptoms [patients] | Changes during baseline and intervention period (measured regularly for 12 weeks)
  The Hospital Anxiety and Depression Scale (HAD) will be used to measure anxiety and depressive symptoms. All items are scored on a 4-point scale.
Quality in psychiatric care [patients] | Changes during baseline and intervention period (measured regularly for 12 weeks)
  The QPC-IP measures quality of care on 30 items using a 4-point scale.
Stress of Conscience [staff] | Changes during baseline and intervention period (measured regularly for 12 weeks)
  The Stress of Conscience Questionnaire (SCQ) will be used to measure the frequencies of stressful situations and the degree to which these lead to stress of conscience among staff.
Quality of care [staff] | Changes during baseline and intervention period (measured regularly for 12 weeks)
  The Quality in Psychiatric Care- Inpatient Staff (QPC-IPS) questionnaire will be used to measure quality of care.
Physical activity [patients and staff] | Changes in physical activity between baseline and intervention
  An electronic device measuring physical activity will be carried by participants during one week before and after rebuilding the ward.

CONTACTS AND LOCATIONS:
Overall Officials: Britt-Marie Lindgren, Principal Investigator — Umeå University
Locations (1):
- Umeå university, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lindgren BM, Molin J, Lundstrom M, Stromback M, Salander Renberg E, Ringner A. Does a new spatial design in psychiatric inpatient care influence patients' and staff's perception of their care/working environment? A study protocol of a pilot study using a single-system experimental design. Pilot Feasibility Stud. 2018 Dec 26;4:191. doi: 10.1186/s40814-018-0383-4. eCollection 2018. PMID 30607254